CLINICAL TRIAL: NCT06347341
Title: GlutN : Randomized, Double-blind, Crossover Clinical Trial to Confirm the Role of Gluten in Non-celiac Gluten Sensitivity
Acronym: GLUTN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient recruitment
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other); UCA (UFR de Médecine et UFR Pharmacie) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2019-A02014-53
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: The Objective is to Confirm the Role of Gluten in Triggering the Digestive and Extradigestive Symptoms of NCGS

STUDY DESIGN:
Intervention Model Description: Prospective, crossover, randomized, double-blind clinical study comparing a gluten-containing diet to a gluten-free diet.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: Clinical study comparing a gluten-containing diet to a gluten-free diet — The study includes a basal period of 2 weeks, 2 test periods of a maximum duration of 1 week and a wash-out period of 2 to 3 weeks.

SUMMARY:
For 25 years, non-celiac gluten sensitivity (NCGS) has been the subject of very prolific and confusing scientific literature. This clinical entity is defined by the appearance of digestive and extradigestive symptoms in the hours/days following the consumption of foods containing gluten, in the absence of celiac disease (CD) and wheat allergy (WA). The physiopathological mechanisms, neither allergic or autoimmune, remain poorly defined and no The main objective of the study was to demonstrate the role of gluten in triggering digestive symptoms and extradigestive products from the NCGS. The secondary objectives were to identify the pathophysiological mechanisms and diagnostic marker(s).usable diagnostic marker in the clinic has not yet been identified.

DETAILED DESCRIPTION:
Twenty patients with possible NCGS on clinical examination and after elimination of CD and AB were included in a study monocentric, randomized, double-blind and crossover design, comparing a gluten-containing diet (RAG) to a gluten-free diet (RSG). The inclusion visit included a specific questioning about digestive and extradigestive symptoms triggered by the consumption of foods with gluten, personal and family history of autoimmune disease, allergy, atopic condition. A dietary consultation made it possible to specify the strict and controlled RSG in FODMAPs (basal diet - RB) to be maintained throughout the 6 weeks of study. After an initial period (PI) of 2 weeks with this RB, patients added for 1 week either foods with gluten (8 g of gluten/d - RAG) or gluten-free foods (RSG) (test periods - PT), the 2 PT being separated by a wash-out period (PWO) of 2 to 3 weeks. Digestive and extradigestive symptoms were assessed by the modified Gastrointestinal Symptom Rating Scale (GSRS) using a 7-point Likert scale (1: absent - 7: very severe), at the end of each week of IP and PWO ( D7 and D14) and every day of each PT. If the symptoms were too severe during PT (i.e. sides of 7), the patient was allowed to stop after a minimum of 72 hours of consumption. For the study of markers of inflammation, immunity, intestinal permeability and metabolomic analyses, blood and urine samples were taken at inclusion and at the end of each PT (or at the end premature). The primary endpoint was the difference in GSRS score at the end of the 2 PTs. Statistical analyzes were carried out using mixed models for a crossover design taking into account subject, diet, period, order and sequence effects and their interactions.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman, aged over 18, suspected of gluten sensitivity defined by the existence of digestive and extradigestive symptoms when consuming foods containing gluten, disappearing in the absence of gluten consumption.
* Patient able to provide informed consent to participate in research.
* Patient covered by a Social Security plan.

Exclusion Criteria:

* - Weight < 45 kg
* Celiac disease: presence of anti-tissue transglutaminase and/or anti-endomysium autoantibodies and/or villous atrophy found on duodenal biopsies.
* Wheat allergy: presence of IgE specific to wheat and/or positivity of prick tests and/or patch tests.
* Presence of another food intolerance/sensitivity, in particular to vegetables and fruits rich in FODMAPs, excluding lactose intolerance (extremely common, 30 to 50% of the French population).
* Presence only of digestive symptoms, without extradigestive symptoms, when consuming foods containing gluten.
* Impossibility of eliminating celiac disease: HLA DQ2 or DQ8 patient, for whom we do not have a dosage of anti-transglutaminase/anti-endomysium antibodies and/or duodenal histology on a normal diet containing gluten.
* Current special diet: vegetarian diet except ovo-lactovegetarian or ovo-lacto-pescovegetarian (i.e. pesco-vegetarian diet, vegan/vegan diet, macrobiotic diet, etc.), Paleolithic diet, etc.
* Pregnant or breastfeeding women.
* Treatment in progress or for less than two months with NSAIDs, corticosteroids, antibiotics, probiotics, food supplement (glutamine, omega3, antioxidants, etc.) and any other treatment likely to interfere with the study (left to the discretion of the patient). 'investigator).
* Current treatment or for less than 18 months with immunosuppressants, chemotherapy.
* History of digestive surgical intervention (except cholecystectomy and appendectomy).
* Any infectious or inflammatory pathology in progress or less than a month old and any other pathology likely to interfere with the protocol (left to the discretion of the investigator).
* Individual under guardianship, curatorship or legal protection, or deprived of freedoms.
* Participation in another clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-03-24 (Actual)

PRIMARY OUTCOMES:
The main objective of the study is to confirm the role of gluten in triggering the digestive and extradigestive symptoms of NCGS. | The patient must complete the questionnaire at the end of each week of the basal period (lasting 2 weeks) and the wash-out period (lasting 2 to 3 weeks) and every day of each test period.
  The GSRS includes 15 digestive symptoms and 9 extradigestive symptoms, rated on a LIKERT scale from 1 (no symptoms) to 7 (extremely severe symptoms).

CONTACTS AND LOCATIONS:
Overall Officials: corinne Bouteloup, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Estaing, Clermont-Ferrand, France